CLINICAL TRIAL: NCT01035242
Title: "Association Splitting" Compared With Cognitive Remediation (CR) in Obsessive-compulsive Disorder (OCD): a Randomized Controlled Trial
Brief Title: "Association Splitting" in Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JE 540/3-1
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; obsessions; cognitive
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Obsessive Behavior | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- "association splitting" (Experimental): Association splitting (6 sessions) delivered by psychologists.
  Interventions: Behavioral: "association splitting"
- cognitive remediation (Active Comparator): CogPack training(6 sessions) delivered by either psychologists or psychology students at an advanced master level.
  Interventions: Behavioral: cognitive remediation

INTERVENTIONS:
Behavioral: "association splitting" — "Association splitting" is a cognitive intervention which aims at reducing obsessive thoughts. Association splitting is based on the so called fan effect (Anderson, 1974) and aims at reducing the strength of obsessive cognitions. For this purpose core intrusive thoughts are identified with the patient (such as "cancer - illness") and the patient is encouraged to find non-OCD associations that are (semantically or phonologically) related to the OCD cognition (such as "cancer - (zodiac) sign", "cancer - great crab"). To strengthen the novel connections, these associations are elaborated by the use of pictures, music, or smells. By enhancing OC-unrelated associations it is assumed that the influence of OC-related concepts is weakened.
  Arms: "association splitting"
Behavioral: cognitive remediation — Computerized cognitive remediation (CogPack training). A fixed sequence is administered, which covers a wide range of neuropsychological exercises involving memory, reasoning, selective attention and psychomotor speed. The difficulty level for each patient is adapted automatically depending on to the subject's performance on prior exercises. At the end of each session, the patient receives individual feedback on his or her performance. To match with association splitting, six sessions are administered. Each session lasts approximately 45-60 minutes.
  Arms: cognitive remediation

SUMMARY:
Over a period of 3 weeks, association splitting is compared to cognitive remediation (CogPack training) as an add-on intervention to cognitive-behavioral therapy (CBT). Blind to treatment assignment, both groups are assessed before intervention and eight weeks as well as six months later with the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), the Obsessive-Compulsive Inventory (OCI-R) and cognitive tests. OCD severity as measured by the Y-BOCS total score serves as the primary outcome parameter. It is assumed that association splitting will improve OCD severity to a greater extent than cognitive remediation.

DETAILED DESCRIPTION:
Association splitting is a new cognitive technique which aims at reducing obsessive thoughts. It draws upon the so-called "fan effect" of associative priming. Transposing this principle to the treatment of obsessive-compulsive disorder (OCD), we hypothesized that the sprouting of new and the strengthening of existing neutral associations to core OCD cognitions will reduce their fear-evoking properties by depriving the chain of OCD-related cognitions of associative strength. Patients with OCD are randomly allocated to either associations splitting (AS) or cognitive remediation (CogPack training). Blind to treatment assignment, both groups are assessed before intervention and eight weeks as well as six months later with the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), the Obsessive-Compulsive Inventory (OCI-R) and cognitive tests. OCD severity derived from the Y-BOCS and the OCI-R serves as the main outcome parameters. We also explore if AS changes the OCD-related semantic networks with cognitive tasks. It is assumed that association splitting will improve OCD severity to a greater extent than CogPack training.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive-Compulsive Disorder (OCD) with an Y-BOCS obsession subscore ≥ 8

Exclusion Criteria:

* intellectual disability (IQ < 70); unable to provide informed consent; severe neurological illness, psychotic symptoms or substance dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Total score of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 8 weeks, 6 months

SECONDARY OUTCOMES:
Obsession subscore of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) and the total score of the Obsessive-Compulsive Inventory (OCI-R) | 8 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lena Jelinek, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Steffen Moritz, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg Eppendorf, Hamburg, Hamburg, Germany

REFERENCES:
- [Result] Jelinek L, Hauschildt M, Hottenrott B, Kellner M, Moritz S. Further evidence for biased semantic networks in obsessive-compulsive disorder (OCD): when knives are no longer associated with buttering bread but only with stabbing people. J Behav Ther Exp Psychiatry. 2014 Dec;45(4):427-34. doi: 10.1016/j.jbtep.2014.05.002. Epub 2014 May 24. PMID 24929782